CLINICAL TRIAL: NCT03489564
Title: The Effect of Physical Activity on in Vivo and in Vitro Mitochondrial Capacity in Pregnant Women
Brief Title: Mitochondrial Capacity in Pregnant Women
Acronym: Mito Moms
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Associate Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2017-065
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy Related; Physical Activity
Keywords: Pregnancy; Mitochondrial metabolism; Placenta
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Placental biospecimens (placenta, umbilical cord, cord blood). Leg muscle tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active: Physically active will be defined by self-report and confirmed by step counts >8,000 per day from activity monitoring.
  Interventions: Behavioral: Active
- Sedentary: Sedentary lifestyle will be defined by self-report and confirmed by step counts <5,000 per day from activity monitoring.
  Interventions: Behavioral: Sedentary

INTERVENTIONS:
Behavioral: Active — No behavioral intervention included but the exposure is level of physical activity. Individuals in the Active group will be categorized by their own routine physical activity levels.
  Groups: Active
Behavioral: Sedentary — No behavioral intervention included but the exposure is level of physical activity. Individuals in the Sedentary group will be categorized by their own routine physical activity levels.
  Groups: Sedentary

SUMMARY:
This Pilot & Feasibility study will test the hypothesis that pregnant women who are more active will have better functioning mitochondria in vivo (higher ATPmax, via 31P-MRS), which will be positively related to maternal and infant mitochondrial function in vitro (higher oxygen consumption rates in primary myotubes and umbilical cord derived mesenchymal stem cells, respectively). Twenty pregnant women (10 active and 10 sedentary) will be recruited in the first trimester of pregnancy determined from self-reported physical activity and assessment by activity monitors. Placental biospecimens will be collected during delivery for other molecular mitochondrial analyses.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female
* BMI between 18.5 kg/m2 and 30.0 kg/m2 prior to the current pregnancy (determined by self report and confirmation of pregravid BMI of the index pregnancy from the prenatal record)
* Medically cleared for participation in the study by primary care obstetrician or midwife
* Medically cleared for participation by the Medical Investigator
* Medical record release (prenatal record, hospital delivery record) for study staff to access information in the medical record related to the current and if applicable, the prior pregnancy.

Exclusion Criteria:

* Risk of early delivery (eg. history of preterm birth, spontaneous abortion, evidence of gestational hypertension (SBP >160 mmHg & DBP >110 mmHg) or pre-eclampsia in the current pregnancy)
* History of intrauterine growth-restriction
* Persistent second- or third-trimester bleeding
* Placenta previa after 26 weeks gestation
* Incompetent cervix or cerclage
* Severe anemia
* High-order pregnancy (e.g. triplets)
* Family history of diabetes
* Heart or lung disease
* HIV or AIDS (self-reported)
* Individuals with contraindication to magnetic resonance spectroscopy such as having magnetic metallic objects in their body
* Unwillingness for placental biospecimens to be collected at delivery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Healthy women that are classified as either physically active or sedentary in early pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Infant in vitro mitochondrial capacity (by oxygen consumption rate) | 1 day
  Infant in vitro mitochondrial capacity measured by oxygen consumption rates in umbilical cord derived mesenchymal stem cells at delivery

SECONDARY OUTCOMES:
Relationship between in vivo mitochondrial capacity and infant in vitro mitochondrial capacity (by oxygen consumption rates) | About 20 weeks
  Relationship between in vivo and in vitro mitochondrial capacity will be measured with in vivo mitochondrial capacity measured by 31P-MRS and infant in vitro mitochondrial capacity measured by oxygen consumption rates in umbilical cord derived mesenchymal stem cells
Relationship between in vivo mitochondrial capacity and maternal in vitro mitochondrial capacity (by oxygen consumption rate) | About 15 weeks
  Relationship between in vivo and in vitro mitochondrial capacity will be measured with in vivo mitochondrial capacity measured by 31P-MRS and maternal in vitro mitochondrial capacity measured by oxygen consumption rates in maternal primary myotubes

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pennington Biomedical Research Center website description and webscreener survey — http://www.pbrc.edu/clinical-trials/?studyid=260